CLINICAL TRIAL: NCT06964828
Title: Proof of Concept, Randomized, Controlled, and Crossover Study, to Assess the Effectiveness of Two Types of Compression Garments (Flat vs Circular Knitted) in the Maintenance Treatment of Patients With Lipedema
Brief Title: Proof of Concept, Randomized, and Crossover Study, to Assess the Effectiveness of Two Types of Compression Garments in Lipedema
Acronym: LipeGar
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Isabel Forner-Cordero, MD, PhD (Other)
Collaborators: Hospital Provincial de Castellon (Other); Hospital Arnau de Vilanova (Other)
Responsible Party: Sponsor-Investigator, Isabel Forner-Cordero, MD, PhD, MD, PhD, Specialist in Physical Medicine and Rehabilitation, Associate professor of University of Valencia, Instituto de Investigacion Sanitaria La Fe
Organization: Instituto de Investigacion Sanitaria La Fe (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LipeGar
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Lipedema
Keywords: Lipedema; Compression garments; Maintenance treatment
MeSH Terms: conditions — Lipedema

STUDY DESIGN:
Intervention Model Description: Patients meeting the inclusion criteria will be randomized to either continue wearing a compression garment with circular fabric or switch to a compression garment with flat fabric, both for 6 months. At 6 months, the study goals will be evaluated, and a simple crossover will occur. Patients will switch to the other type of garment for another 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Circular-knitted compression garments (Active Comparator): The patient will continue using a compression garment with the same fabric she was wearing before inclusion (circular knitted pantyhose in class 2)
  Interventions: Device: Flat-knitted compression garment
- Flat-knitted compression garments (Experimental): The patient will change to a flat-knitted pantyhose in class 2 for 6 months
  Interventions: Device: Flat-knitted compression garment

INTERVENTIONS:
Device: Flat-knitted compression garment — Flat knitted compression garments
  Other Names: Circular-knitted compression garment

SUMMARY:
The goal of this prospective randomized crossover experimental study is to assess the effectiveness and tolerance of circular and flat fabric garments in stabilizing lower-limb volume in lipedema. It will assess the effectiveness of the garments and determine any differences between both types of hosiery currently used in routine clinical practice. Participants will be prescribed either circular or flat-knitted pantyhose and wear them daily for 6 months. After 6 months, they will change the type of garment.

DETAILED DESCRIPTION:
Lipedema, described by Allen and Hines in 1940, is a syndrome characterized by painful edema in the lower limbs associated with a frequent occurrence of bruises. It mainly affects women and is usually symmetrical.

The management of patients depends on the stage and the presence of edema. In the maintenance phase, the goal is to prevent edema recurrence to avoid an increase in fat deposition in the lower limbs through the use of compression garments.

Currently, there are no guidelines for prescribing compression garments for patients with lipedema regarding the type of garment, fabric, or compression level. Therefore, the prescription by lymphologists is empirical and based on experience.

This study, the first of its kind, aims to assess the effectiveness and tolerance of circular and flat fabric garments in stabilizing the volume of the lower limbs and improving or stabilizing the signs and symptoms of patients with lipedema. The study also aims to determine if there are differences between the two types of garments currently used in routine clinical practice.

In order to provide scientific knowledge to guide these decisions, a prospective randomized crossover experimental study is proposed in patients with lipedema type III, stages 1 and 2, undergoing maintenance treatment with circular compression stockings for a minimum of 6 months. Patients meeting inclusion criteria will be randomized to continue receiving a compression garment with the same circular fabric they were wearing or alternatively switch to a compression garment with flat fabric, both for 6 months.

After 6 months, the study goals will be evaluated, and a simple crossover will be performed, switching to the other type of garment for another 6 months. In other words, patients wearing circular fabric garments will change to flat fabric compression garments and vice versa. At the end of the subsequent 6 months, the study goals will be reassessed once more.

To assess the study goals, we will record several variables related to:

* The effectiveness of circular and flat fabric garments
* Patient satisfaction with the garments
* Compliance with garment use
* Patient complaints about the garments

Therefore, patients will be recieve a follow-up visit at 6 months from the baseline assessment and at 6 months after crossover treatment. Garment usage will be assessed through automated calls every 2 weeks during the whole follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of lipedema: increased lowe-limb volume, disproportion between upper and lower body, and pain.
* Lipedema type III stages 1 or 2.
* Negative pitting sign.
* In maintenance treatment phase with a class II circular-knitted compression garment for at least 6 months.
* Adequate compliance with compression garments (worn during the day, except during personal hygiene and water-related activities).
* Written informed consent to participate.

Exclusion Criteria:

* Lipedema with fatty lobulations.
* Body Mass Index (BMI) ≥ 30 kg/m2.
* Waist-to-Height Ratio > 0.53.
* Pregnancy.
* Renal, hepatic, or cardiac insufficiency.
* Thrombosis in the lower extremities.
* Infection in the lower extremities.
* Active oncological process.
* Current treatment with corticosteroids and other medications that promote fluid retention.
* Inability to read the Patient Information Form (HIP) and/or provide consent to participate in the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Volume Change (PVC) | at the 6th and 12th month of treatment
  The Percentage of Volume Change (PVC) at the 6th and 12th month of treatment is calculated using the following mathematical formula:
  PVC = [ (Baseline volume- final volume)/ baseline volume] x 100
  Where:
  * Baseline is the reference volume at the beginning of the treatment.
  * Final Volume is the volume at the end of the treatment period (either at the 6th or 12th month).
  This calculation provides the percentage change in volume of the lower limbs over the course of the treatment period compared to the initial volume.
  We consider maintenance treatment is successful when the Percentage of Volume Change (PVC) is <10% after 6 or 12 months of treatment, relative to the study's baseline. We define disease progression when the PVC is >10% at 6 or 12 months, relative to the study's baseline.

SECONDARY OUTCOMES:
Pain intensity | at the 6th and 12th month of treatment
  Pain in lower limbs: visual analogue scale (VAS). Scores range from 0 (absent) to 10 (worst possible).
Heaviness | at the 6th and 12th month of treatment
  Perceived heaviness in lower limbs: visual analogue scale (VAS). Scores range from 0 (absent) to 10 (worst possible).
Numbness | at the 6th and 12th month of treatment
  Numbness in lower limbs: visual analogue scale (VAS). Scores range from 0 (absent) to 10 (worst possible).
Characteristics of pain | at the 6th and 12th month of treatment
  Location and type of sensation.
Compliance | at the 6th and 12th months of treatment
  Number of hours per day and days per week, wearing the compression garments
Reported Quality of Life | at the 6th and 12th months of treatment
  LYMQOL (Lymphedema Quality of Life) questionnaire. Individual item scores range from 0 (least impact in quality of life or QOL) to 4 (maximum impact in QOL). Total scores may be calculated as a mean of all individual answers or as a percentage of the maximum possible score. The last question regarding overall quality of life is measured using the visual analogue scale (VAS) ranging from 0 (worst possible QOL) to 10 (best possible QOL).
Pressure pain threshold | at baseline, 6th and 12 th months.
  Pressure pain threshold (PPT) will be assessed at the thigh using an algometer. Units: Newtons (N).

CONTACTS AND LOCATIONS:
Overall Officials: ISABEL FORNER-CORDERO, MD, PhD, Principal Investigator — Hospital Universitario La Fe
Locations (1):
- Hospital Universitari i Politecnic La Fe, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michelini S, Chiurazzi P, Marino V, Dell'Orco D, Manara E, Baglivo M, Fiorentino A, Maltese PE, Pinelli M, Herbst KL, Dautaj A, Bertelli M. Aldo-Keto Reductase 1C1 (AKR1C1) as the First Mutated Gene in a Family with Nonsyndromic Primary Lipedema. Int J Mol Sci. 2020 Aug 29;21(17):6264. doi: 10.3390/ijms21176264. PMID 32872468
- [Background] Ghods M, Georgiou I, Schmidt J, Kruppa P. Disease progression and comorbidities in lipedema patients: A 10-year retrospective analysis. Dermatol Ther. 2020 Nov;33(6):e14534. doi: 10.1111/dth.14534. Epub 2020 Nov 22. PMID 33184945
- [Background] Herbst KL, Mirkovskaya L, Bharhagava A, Chava Y, Te CHT. Lipedema fat and signs and symptoms of illness, increase with advancing stage. Archives of Medicine. 2015; 7(4): 1-8.
- [Background] Kumar B, Lenert P. Joint Hypermobility Syndrome: Recognizing a Commonly Overlooked Cause of Chronic Pain. Am J Med. 2017 Jun;130(6):640-647. doi: 10.1016/j.amjmed.2017.02.013. Epub 2017 Mar 10. PMID 28286166
- [Background] Forner-Cordero I, Muñoz-Langa J, Vázquez-Díez J. Lipedema patients have a high prevalence of joint hypermobility. ISL XXVII WORLD CONGRESS 2019, International Society of Lymphology, Buenos Aires (Argentina), September 23-28, 2019.
- [Background] WOLD LE, HINES EA Jr, ALLEN EV. Lipedema of the legs; a syndrome characterized by fat legs and edema. Ann Intern Med. 1951 May;34(5):1243-50. doi: 10.7326/0003-4819-34-5-1243. No abstract available. PMID 14830102
- [Background] Herbst KL. Rare adipose disorders (RADs) masquerading as obesity. Acta Pharmacol Sin. 2012 Feb;33(2):155-72. doi: 10.1038/aps.2011.153. PMID 22301856
- [Background] Schmeller W, Meier-Vollrath I. Das Lipodem: neue Möglichkeiten der Therapie. Schweiz Med Forum. 2007;7:150-155.
- [Background] Halk AB, Damstra RJ. First Dutch guidelines on lipedema using the international classification of functioning, disability and health. Phlebology. 2017 Apr;32(3):152-159. doi: 10.1177/0268355516639421. Epub 2016 Jul 9. PMID 27075680
- [Background] Lontok E, Briggs L, Donlan M, Kin Y, Mosley E, Riley EAU, Stevens M. Lipedema. A giving smarter guide. Milken Institute center for strategic philanthropy. 2017.
- [Background] Hardy D, Williams A. Best practice guidelines for the management of lipoedema. Br J Community Nurs. 2017 Oct 1;22(Sup10):S44-S48. doi: 10.12968/bjcn.2017.22.Sup10.S44. No abstract available. PMID 28961048
- [Background] Dayan E, Kim JN, Smith ML, editors. Lipedema - The disease they call FAT: An overview for clinicians. Boston, MA: Lipedema Simplified Publications, The Friedman Center for Lymphedema Research and Treatment at The Center for Advanced Medicine at Northwell Health in collaboration with Lymphatic Education & Research Network (LE&RN); 2017.
- [Background] Nemes A, Kormanyos A, Domsik P, Kalapos A, Kemeny L, Szolnoky G. The impact of lower body compression garment on left ventricular rotational mechanics in patients with lipedema-Insights from the three-dimensional speckle tracking echocardiographic MAGYAR-Path Study. Clin Obes. 2020 Oct;10(5):e12380. doi: 10.1111/cob.12380. Epub 2020 Jun 23. PMID 32573965
- [Background] Forner-Cordero I, Tortosa-Soriano G, Alabajos-Cea A, Ponce-Garrido AB, Muñoz-Langa J. Effect of compression alone or combined with exercise in patients with lipedema. A pilot study. In: Abstracts of the 42nd European Society of Lymphology Congress. Eur J Lymphol Relat Probl. 2016; 28(74): 70.
- [Background] Reich-Schupke S, Schmeller W, Brauer WJ, Cornely ME, Faerber G, Ludwig M, Lulay G, Miller A, Rapprich S, Richter DF, Schacht V, Schrader K, Stucker M, Ure C. S1 guidelines: Lipedema. J Dtsch Dermatol Ges. 2017 Jul;15(7):758-767. doi: 10.1111/ddg.13036. PMID 28677175
- [Background] Flour M, Clark M, Partsch H, Mosti G, Uhl JF, Chauveau M, Cros F, Gelade P, Bender D, Andriessen A, Schuren J, Cornu-Thenard A, Arkans E, Milic D, Benigni JP, Damstra R, Szolnoky G, Schingale F. Dogmas and controversies in compression therapy: report of an International Compression Club (ICC) meeting, Brussels, May 2011. Int Wound J. 2013 Oct;10(5):516-26. doi: 10.1111/j.1742-481X.2012.01009.x. Epub 2012 Jun 21. PMID 22716023
- [Background] Forner-Cordero I, Szolnoky G, Forner-Cordero A, Kemeny L. Lipedema: an overview of its clinical manifestations, diagnosis and treatment of the disproportional fatty deposition syndrome - systematic review. Clin Obes. 2012 Jun;2(3-4):86-95. doi: 10.1111/j.1758-8111.2012.00045.x. Epub 2012 Aug 3. PMID 25586162
- [Background] Forner-Cordero I, Perez-Pomares MV, Forner A, Ponce-Garrido AB, Munoz-Langa J. Prevalence of clinical manifestations and orthopedic alterations in patients with lipedema: A prospective cohort study. Lymphology. 2021;54(4):170-181. PMID 35073621
- [Background] Forner-Cordero I, Forner-Cordero A, Szolnoky G. Update in the management of lipedema. Int Angiol. 2021 Aug;40(4):345-357. doi: 10.23736/S0392-9590.21.04604-6. Epub 2021 Apr 19. PMID 33870676
- [Background] Paling I, Macintyre L. Survey of lipoedema symptoms and experience with compression garments. Br J Community Nurs. 2020 Apr 1;25(Sup4):S17-S22. doi: 10.12968/bjcn.2020.25.Sup4.S17. PMID 32271105
- [Background] Kurz I. Textbook of Dr. Vodder's manual lymph drainage. In: Harris RS, editors. Therapy. 2nd ed. Heidelberg (Germany): Karl S. Haug Publishers; 1989
- [Background] Chen YW, Tsai HJ, Hung HC, Tsauo JY. Reliability study of measurements for lymphedema in breast cancer patients. Am J Phys Med Rehabil. 2008 Jan;87(1):33-8. doi: 10.1097/PHM.0b013e31815b6199. PMID 17993983
- [Background] Meijer RS, Rietman JS, Geertzen JH, Bosmans JC, Dijkstra PU. Validity and intra- and interobserver reliability of an indirect volume measurements in patients with upper extremity lymphedema. Lymphology. 2004 Sep;37(3):127-33. PMID 15560108
- [Background] Deltombe T, Jamart J, Recloux S, Legrand C, Vandenbroeck N, Theys S, Hanson P. Reliability and limits of agreement of circumferential, water displacement, and optoelectronic volumetry in the measurement of upper limb lymphedema. Lymphology. 2007 Mar;40(1):26-34. PMID 17539462
- [Background] Belgrado JP, Bracale P, Bates J, Röh N, Rosiello R, Cangiano A, et al. Lymphoedema: what can be measured and how… overview. Eur J Lymphol Relat Probl. 2010; 21(61):3-9
- [Background] Cuello-Villaverde E, Forner-Cordero I, Forner-Cordero A. Linfedema: métodos de medición y criterios diagnósticos. Rehabilitación (Madr). 2010;44:21-8.